CLINICAL TRIAL: NCT03632109
Title: Gentamicin for Pharyngeal Gonorrhea - A Demonstration Study
Brief Title: Gent for Pharyngeal Gonorrhea (GC)
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Efficacy
Sponsor: University of Washington (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Lindley Barbee, Assistant Professor, School of Medicine: Department of Medicine: Allergy and Infectious Diseases, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003878; K23AI113185 (NIH)
Record Dates: First submitted 2018-07-03; First posted 2018-08-15 (Actual); Results first posted 2020-08-10 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-07

CONDITIONS: Pharyngeal Gonococcal Infection
Keywords: gonorrhea; pharynx; treatment; gentamicin
MeSH Terms: conditions — Gonorrhea | interventions — Gentamicins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental): Men who have sex with men (MSM) with pharyngeal gonorrhea will be treated with 360mg intramuscular gentamicin x 1.
  Interventions: Drug: gentamicin 360mg IM

INTERVENTIONS:
Drug: gentamicin 360mg IM — 360mg IM of gentamicin

SUMMARY:
The Centers for Disease Control and Prevention has identified antimicrobial-resistant (AMR) Neisseria gonorrhoeae (NG) as one of the nation's top three urgent AMR threats. Since the advent of antibiotics in the 1930s, NG has developed resistance to every first-line antibiotic. Parenteral third-generation cephalosporins are now the only class of drug with consistent efficacy against NG. New therapies are urgently needed. Although some novel antimicrobials are under development, reevaluating older drugs is another option for quickly identifying additional treatments for gonorrhea. We propose a demonstration study to test a single dose of gentamicin for the treatment of pharyngeal gonorrhea. We chose to focus on pharyngeal gonorrhea because these infections are common, play an important role in fostering gonococcal resistance, and are harder to eradicate than genital infections. Although gentamicin is 91% efficacious for genital NG, its efficacy at the pharynx may be less since streptomycin, another aminoglycoside previously used to treat gonorrhea, was not effective for pharyngeal NG. It is unknown if streptomycin's poor efficacy is indicative of limitations of aminoglycosides as a class. We plan to enroll 60 men who have sex with men in a demonstration study to be conducted at the Seattle & King County STD Clinic to test the efficacy of 360 mg of gentamicin given intramuscularly for pharyngeal gonorrhea. Secondary objectives include determining the ideal pharmacodynamic criterion (comparing in vitro minimal inhibitory concentrations (MIC) of NG to peak gentamicin serum levels), estimating resistance induction among treatment failures, and assessing the tolerability of 360 mg of IM gentamicin.

Objectives

The proposed study aims to evaluate the efficacy of a single intramuscular (IM) dose of gentamicin in the treatment of pharyngeal gonorrhea. Secondary objectives include documenting the efficacy stratified by minimal inhibitory concentration (MIC) compared with the gentamicin peak level in order to estimate a pharmacodynamic criterion. We will also attempt to determine whether gentamicin monotherapy induces antimicrobial resistance among treatment failures. Lastly, we will evaluate the tolerability of 360 mg of IM gentamicin, stratified by subject weight (i.e. weight based dosing). The specific aims are:

1. Determine the proportion of persons whose pharyngeal gonococcal infections are cured with a single dose of 360mg gentamicin intramuscularly alone.
2. Evaluate the renal safety and tolerability of 360mg IM of gentamicin.
3. Document mean peak gentamicin levels following 360mg IM of gentamicin stratified by weight.
4. Estimate the best pharmacodynamics criterion (i.e. peak/MIC ratio) for pharyngeal gonorrhea treated with gentamicin using individual and mean peak gentamicin levels and NG isolate MIC.
5. Among treatment failures, conduct exploratory analyses comparing pre- and post-treatment MIC for evidence of induced resistance.

ELIGIBILITY:
Inclusion Criteria:

* Persons diagnosed with pharyngeal gonorrhea who are not yet treated

Exclusion Criteria:

* Age less than 16 years
* Receipt of antibiotics in ≤30 days
* Known allergy to any aminoglycoside
* History of renal disease (including diagnosis of solitary kidney, chronic renal insufficiency, renal cell carcinoma etc),
* Use of concurrent nephrotoxic drugs or muscle relaxants
* History of diabetes
* History of hearing loss or tinnitus
* Concurrent infection with syphilis or chlamydia
* Pregnancy and/or nursing
* Unable to return for a follow-up visit 4-7 days (+/- 1 day).
* Study team's discretion

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2019-03-12 (Actual); Study Completion 2019-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindley A Barbee, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- Public Health -- Seattle & King County STD Clinic, Seattle, Washington, United States

REFERENCES:
- [Derived] Barbee LA, Soge OO, Morgan J, Leclair A, Bass T, Werth BJ, Hughes JP, Golden MR. Gentamicin Alone Is Inadequate to Eradicate Neisseria Gonorrhoeae From the Pharynx. Clin Infect Dis. 2020 Nov 5;71(8):1877-1882. doi: 10.1093/cid/ciz1109. PMID 31712813

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm: Pharyngeal Gonorrhea
Period: Overall Study
Arm/Group | Single Arm
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 13
Age, Continuous [Mean (Full Range); unit: years] | 29.3 [21 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13
Weight (kg) [Mean (Full Range); unit: kg] | 86.4 [53 to 133]
Height (in) [Mean (Full Range); unit: in] | 70.9 [68 to 76]
BMI (kg/m2) [Mean (Full Range); unit: kg/m^2] | 26.6 [17.9 to 43.4]
Baseline Creatinine [Mean (Full Range); unit: mg/dL] | 0.86 [0.74 to 1.05]
PrEP Status (Taking HIV PrEP) [Count of Participants; unit: Participants] | 8
Number of oral sex partners in the last 2 months [Mean (Full Range); unit: reported sex partners] | 4.2 [0 to 10]

OUTCOME MEASURES:

1. Primary Outcome: Cure Rate Defined as the Percentage of Persons With Pharyngeal Gonorrhea Treated With Gentamicin 360mg IM Who Have a Negative Culture 4-7 Days Following Treatment
Description: Negative Pharyngeal Culture
Time Frame: 4-7 days (+/- 1 day) after treatment
Population: Positive culture at enrollment and returned for test of cure, or negative culture at enrollment but positive culture at test of cure
Measure: Count of Participants; unit: Participants
Groups:
- Pharyngeal Gonorrhea: Evaluable Population
Arm/Group | Pharyngeal Gonorrhea
Number analyzed (Participants) | 10
Participants | 2

2. Secondary Outcome: Renal Safety
Description: Measured by a percent change in serum creatinine from baseline to test of cure (4-7 days following treatment)
Time Frame: 4-7 days (+/- 1 day) after treatment
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Single Arm
Number analyzed (Participants) | 13
percent change | 5.2 [0.20 to 10.1]

3. Secondary Outcome: Tolerability of the Injection Gentamicin 360mg IM x 1
Description: Participant reported pain scale, with 1 being little to no pain, and 10 being the worst pain ever.
Time Frame: 4-7 days (+/- 1 day) after treatment
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 13
score on a scale | 2 [1 to 7]

4. Secondary Outcome: Peak Gentamicin Levels
Description: serum gentamicin concentration
Time Frame: at 30, 45, or 60 minutes post dose
Population: 2 participants had missing gentamicin levels
Measure: Mean (Full Range); unit: microgram/mL
Arm/Group | Single Arm
Number analyzed (Participants) | 11
microgram/mL | 21.2 [15 to 30]

5. Secondary Outcome: Gentamicin Minimal Inhibitory Concentration (MIC)
Description: laboratory defined MIC of infecting strain of N. gonorrhoeae at enrollment visit determined by agar dilution
Time Frame: baseline/enrollment visit
Population: 2 participants were culture negative at enrollment
Measure: Mean (Full Range); unit: microgram/mL
Arm/Group | Single Arm
Number analyzed (Participants) | 11
microgram/mL | 6.9 [4 to 8]

6. Other Pre Specified Outcome: Exploratory Study: Look for Evidence of Induced Resistance
Description: Among treatment failures, compare pre-treatment and post-treatment minimal inhibitory concentrations (MIC)
Time Frame: 4-7 days (+/- 1 day) after treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected at the test of cure visit 4-7 days following dosing.
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 7/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=13)
Headache (Nervous system disorders) | 6
Fatigue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Hearing Changes (Ear and labyrinth disorders) | 1
Urine Changes (Renal and urinary disorders) | 1
Vomiting (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-04): https://cdn.clinicaltrials.gov/large-docs/09/NCT03632109/Prot_SAP_000.pdf